CLINICAL TRIAL: NCT03660124
Title: Deep Brain Stimulation (DBS) for the Treatment of Refractory Alcohol Use Disorder (AUD): Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012-2018
Record Dates: First submitted 2018-08-07; First posted 2018-09-06 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation Treatment (Experimental)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — DBS is a neurosurgical procedure that involves the administration of small amounts of electricity to disrupt abnormal activity of brain structures associated with disease symptoms. It involves inserting thin electrodes into deep brain structures and electrically stimulating them in a controllable and ultimately reversible manner. The electrodes are connected to an internal pulse generator that is implanted in the upper chest region, below the collarbone.

SUMMARY:
This is a phase I, non-blinded, non-randomized, pilot trial for safety and efficacy of DBS for AUD. Patients who meet inclusion and exclusion criteria will be identified and recruited from the practices of Sunnybrook psychiatrists. Five (5) to ten (10) subjects will be enrolled and study duration for each patient will be of one (1) year. Our primary objective is to establish the safety of DBS in a patient population with treatment refractory AUD. In addition to demonstrating safety, our second primary objective will be to evaluate if DBS-targeted nucleus accumbens in alcoholism is efficacious in the treatment-refractory patients with AUD. This will be measured by various outcome measures that will include validated scales to assess addiction and craving behaviours.

ELIGIBILITY:
Inclusion criteria

1. Female or Male patients between age 18-70
2. Diagnosis of alcohol use disorder (AUD) as defined by the Diagnostic and Statistical Manual fifth edition (DSM-5).
3. History of AUD for at least 2 years, with evidence of repeated failure to respond to evidence-based AUD treatments (psychosocial treatments plus pharmacotherapies such as disulfiram, naltrexone and acamprosate).
4. Alcohol Use Disorders Identification Test (AUDIT) Scale Score >8
5. Ability to provide informed consent and comply with all testing, follow-ups and study appointments and protocols

Exclusion criteria

1. Any past or current evidence of psychosis or mania
2. Current suicidal or homicidal ideation
3. Active neurologic disease, such as epilepsy
4. Visible brain damage or atrophy in CT or MRI scan
5. Any contraindication to MRI or positron emission tomography (PET) scanning
6. Likely to relocate or move during the study's one year duration
7. Presence of clinical and/or neurological conditions that may significantly increase the risk of the surgical procedure.
8. Patients with renal dysfunction (GFR<60)
9. Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | 6 months
  Our primary objective is to establish the safety of deep brain stimulation in a patient population with treatment refractory alcohol use disorder. This is an exploratory pilot study. safety will be reported in the form of adverse event collection, and reported for each patient recruited into the study. Infection, hemorrhage, seizure, sensorymotor disturbance, oculomotor disturbance, or worsening on any adjunctive measure scales used will be reported. These will all be reported on a case-by-case basis, and presented descriptively in the publication. (no specific scale will be used).
Change in Alcohol consumption measured with the alcohol timeline followback | 6 months
  The amount of alcohol consumption preoperatively will be compared with the amount of alcohol consumption postoperatively using the alcohol timeline followback method at 6 months (compared to the preoperative baseline). This will be administered by a psychometrist, and reported as average number of standard drinks consumed daily and weekly during the 6 month postoperative period. An increase from preoperative values is considered a worse outcome, and a decrease in number is an improvement.

SECONDARY OUTCOMES:
Alcohol Dependency Scale | 6 months. This scale is scored out of 47, and will be administered by a psychometrist preoperatively and at 6 months postoperatively. Higher scores are considered worse, so a decrease from baseline is an improvement.
  Alcohol Dependency Scale (ADS) will be compared between preoperative baseline and at 6 month follow up.
Alcohol Urge Questionnaire (AUQ) | 6 months
  Alcohol Urge Questionnaire (AUQ) will be compared between preoperative baseline and at 6 month follow up. This scale is scored out of 84, and will be administered by a psychometrist preoperatively and at 6 months postoperatively. Higher scores are considered worse, so a decrease from baseline is an improvement.
Alcohol Use Disorder Identification Test (AUDIT) | 6 months
  Alcohol Use Disorder Identification Test (AUDIT) will be compared between preoperative baseline and at 6 month follow up.
Hamilton Depression Scale (HAMD) | 6 months
  Hamilton Depression Scale (HAMD) will be compared between preoperative baseline and at 6 month follow up.
Beck Depression and Anxiety Inventory (BDI and BAI) | 6 months. Both the BDI and BAI are scored out of 63, with higher scores indicating a worse outcome. They will be administered by a psychometrist.
  Beck Depression and Anxiety Inventory (BDI and BAI) will be compared between preoperative baseline and at 6 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Davidson B, Giacobbe P, George TP, Nestor SM, Rabin JS, Goubran M, Nyman AJ, Baskaran A, Meng Y, Pople CB, Graham SJ, Tam F, Hamani C, Lipsman N. Deep brain stimulation of the nucleus accumbens in the treatment of severe alcohol use disorder: a phase I pilot trial. Mol Psychiatry. 2022 Oct;27(10):3992-4000. doi: 10.1038/s41380-022-01677-6. Epub 2022 Jul 21. PMID 35858989